CLINICAL TRIAL: NCT02863276
Title: Modulating the Stress Response in Diabetes Mellitus Type 2 Patients Undergoing Colon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 230/09
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus Type 2; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensified insulin group (Experimental): Patients undergoing elective colorectal surgery will receive standard anesthesia including epidural analgesia and nutritional support with an intravenous amino acid solution while receiving tight blood glucose control with intensified insulin therapy (blood glucose target<6 mmol*l-1) via an continuous insulin infusion.
  Interventions: Procedure: Intensified insulin therapy
- Control group (No Intervention): Patients undergoing elective colorectal surgery will receive standard anesthesia including epidural analgesia and nutritional support with an intravenous amino acid solution while receiving standard blood glucose control (blood glucose target <10 mmol*l-1) via subcutaneous insulin boluses

INTERVENTIONS:
Procedure: Intensified insulin therapy
  Other Names: continuous insulin infusion
  Arms: Intensified insulin group

SUMMARY:
Background Surgical injury provokes a stress response. These pathways mediated by stress hormones and cytokines cause a catabolic state. The loss of body cell mass may result in prolonged convalescence and increased morbidity. Protein catabolism after colorectal surgery is even more increased in patients with type 2 diabetes mellitus. Epidural blockade, by reducing the intensity of the catabolic response, improves substrate utilization after surgery in non-diabetic patients. This effect is even more pronounced in diabetic patients receiving amino acids.

The aim of the study is to explore the effect of two different protocols to manage blood glucose control on glucose and protein metabolism in patients with type 2 diabetes mellitus undergoing colon surgery and receiving epidural analgesia and perioperative feeding with amino acids. The following hypotheses are tested:

1. Tight perioperative blood glucose control with intensified insulin therapy compared to standard blood glucose control in presence of general anesthesia with epidural analgesia and amino acid infusion would reduce endogenous glucose production and leucine oxidation.
2. Tight blood glucose control and perioperative infusion of amino acids induce a more positive protein balance compared to standard blood glucose control by better oxidative glucose utilization and redirecting amino acids from oxidative to synthetic pathways.

Material and Methods A total of 20 patients with diabetes mellitus type 2 undergoing elective colorectal surgery will be admitted to the study. Patients will be randomly assigned to receive standard blood glucose control (blood glucose target <10 mmol*l-1; control group; cytotoxic T lymphocyte (CTL) group, n=8) or to receive tight blood glucose control with intensified insulin therapy (blood glucose target<6 mmol*l-1; intensified insulin group; II group, n=8). All patients will receive general anesthesia and an epidural catheter for perioperative analgesia. During surgery (intraoperative state) and immediately after surgery (postoperative state) when receiving an amino acid infusion protein and glucose kinetics will be assessed using a stable isotope technique with L-[1-13C]leucine and [6,6-2H2]glucose and circulating concentrations of glucose, glucagon, insulin and cortisol will be measured. The primary endpoints of the study will be protein balance. Sample size is set to ensure at least 80% power at a significance level of 0.05.

DETAILED DESCRIPTION:
see information below

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colorectal surgery for non-metastatic disease
* Type 2 diabetes mellitus with plasma level of glycosylated hemoglobin level (HbA(1c)) less than 10% indicating normal or moderate glycemic control
* Being capable of signing informed consent
* Accepting an epidural catheter for perioperative analgesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status classification system 4 with major cardiac disorders (severe arrhythmias, recent myocardial ischemia (MI), heart failure, uncontrolled hypertension)
* Hepatic disorders (liver failure, jaundice, metastatic disease), renal disorders (acute or chronic renal failure or on dialysis)
* Metabolic disorders (untreated hyperthyroidism, pyrexia, more than 10% weight loss over the preceding three months, plasma albumin concentration < 35g/l)
* Anemia (hemoglobin < 10 g/dl)
* Chemotherapy or radiotherapy during six months before surgery
* Inflammatory bowel disease or other inflammatory condition
* Pregnancy
* Previous spine surgery precluding placement of an epidural catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Postoperative protein balance (leucine) (umol/kg/h) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine and calorimetry towards the end of the 3 hour period

SECONDARY OUTCOMES:
Intraoperative protein metabolism: Rate of appearance of leucine (umol/kg/h) | Intraoperative period: starting with the induction of anesthesia and ending after 3 hours (during surgery)
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine
Intraoperative protein metabolism: endogenous rate of appearance of leucine (umol/kg/h) | Intraoperative period: starting with the induction of anesthesia and ending after 3 hours (during surgery)
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine
Intraoperative glucose metabolism: Endogenous rate of appearance of glucose (umol/kg/min) | Intraoperative period: starting with the induction of anesthesia and ending after 3 hours (during surgery)
  Measured and calculated with a 3-hour stable isotope tracer technique with D-(6,6-2H2)glucose
Intraoperative glucose metabolism: Glucose clearance (ml/kg/min) | Intraoperative period: starting with the induction of anesthesia and ending after 3 hours (during surgery)
  Measured and calculated with a 3-hour stable isotope tracer technique with D-(6,6-2H2)glucose and plasma glucose measurement
Postoperative protein metabolism: Rate of appearance of leucine (umol/kg/h) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine and calorimetry towards the end of the 3 hour period
Postoperative protein metabolism: Endogenous rate of appearance of leucine (umol/kg/h) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine and calorimetry towards the end of the 3 hour period
Postoperative protein metabolism: Leucine oxidation (umol/kg/h) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine and calorimetry towards the end of the 3 hour period
Postoperative protein metabolism: Protein synthesis (leucine) (umol/kg/h) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with L-(1-13C)leucine and calorimetry towards the end of the 3 hour period
Postoperative glucose metabolism: Endogenous rate of appearance of glucose (umol/kg/min) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with D-(6,6-2H2)glucose
Postoperative glucose metabolism: Glucose clearance (ml/kg/min) | Postoperative period: starting with arrival in the postoperative care unit and ending after 3 hours
  Measured and calculated with a 3-hour stable isotope tracer technique with D-(6,6-2H2)glucose and plasma glucose measurement

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kopp Lugli, MD, MSc, Study Chair — University Hospital, Basel, Switzerland